CLINICAL TRIAL: NCT02522884
Title: Tack Optimized Balloon Angioplasty Study for Superficial Femoral and Proximal Popliteal Arteries Using the Tack Endovascular System™
Brief Title: Tack Optimized Balloon Angioplasty Study of the Tack Endovascular System™ in Femoropoliteal Arteries
Acronym: TOBA II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA 0119
Record Dates: First submitted 2015-08-07; First posted 2015-08-13 (Estimated); Results first posted 2019-12-10 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Peripheral Artery Disease
Keywords: Angioplasty; Peripheral Artery Disease; PAD; Lesion; Claudication
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tack Implant (Experimental): Implantation of a Tack using the Intact Vascular Tack Endovascular System for the repair of post angioplasty dissections.
  Interventions: Device: Tack Endovascular System

INTERVENTIONS:
Device: Tack Endovascular System — Repair of post-PTA dissections using the Intact Vascular Tack Endovascular System.
  Other Names: Post-PTA Dissection Repair Implant; Tack Implant; Tack Dissection Repair Device

SUMMARY:
This is a prospective, multi-center, single-arm, non-blinded study designed to investigate the safety and efficacy of the Tack Endovascular System in subjects with post-balloon angioplasty (post-PTA) dissection(s) type(s) A through F in the superficial femoral and proximal popliteal arteries ranging in diameter from 2.5mm to 6.0mm.

ELIGIBILITY:
Inclusion Criteria:

* Subject must meet all of the following inclusion criteria to be eligible for enrollment:

  1. Male or non-pregnant Female ≥ 18 years of age at the time of consent
  2. Female subjects of childbearing potential must have a negative pregnancy test prior to treatment and must use some form of contraception through the duration of the study (abstinence is acceptable)
  3. Target limb requires no additional treatment aside from the target lesion and the iliac artery(ies) during the index procedure
  4. Subject or has been informed of and understands the nature of the study and provides signed informed consent to participate in the study. If the subject possesses the ability to understand and provide informed consent but due to physical inability, the subject cannot sign the Informed Consent Form, an impartial witness may sign on behalf of the subject
  5. Willing to comply with all required follow-up visits
  6. Rutherford Classification 2, 3 or 4
  7. Estimated life expectancy >1 year
  8. Eligible for standard surgical repair, if necessary
  9. Subject is ambulatory (assistive devices such as a cane or walker is acceptable)

Exclusion Criteria:

* Subject must NOT meet any of the following exclusion criteria to be eligible for enrollment:

  1. Rutherford Classification 0, 1, 5 or 6
  2. Is pregnant or refuses to use contraception through the duration of the study
  3. Previous infrainguinal bypass graft in the target limb
  4. Planned amputation on the target limb
  5. Systemic infection or Infection within the target limb and/or immunocompromised
  6. Endovascular or surgical procedure (not including diagnostic procedures) on the target limb within 30 days prior to or within 30 days after the index procedure
  7. Endovascular or surgical procedure (not including diagnostic procedures) on the non-target limb within 14 days prior to the index procedure or planned procedure within 30 days after the index procedure
  8. Prior coronary artery bypass graft (CABG) or percutaneous coronary intervention (PCI) procedure within 30 days prior to the index procedure or planned CABG/PCI within 30 days after the index procedure
  9. Any other previous or planned surgical or endovascular procedure (not including diagnostic procedures) within 14 days prior to or 30 days post index procedure
  10. Planned atherectomy, cryoplasty, stenting or any other treatment (with the exception of a crossing device) of the target lesion other than PTA during the index procedure
  11. Known coagulopathy, hypercoagulable state, bleeding diathesis, other blood disorder, or a platelet count less than 80,000/microliter or greater than 500,000/microliter
  12. Known hypersensitivity or allergy to antiplatelet or anticoagulant therapy
  13. Myocardial infarction within 30 days prior to enrollment
  14. History of stroke within 90 days prior to enrollment
  15. Serum creatinine of >2.5 mg/dL
  16. Requires treatment of tibial or outflow vessels at the index procedure, which include the P2 and P3 segments of the popliteal artery and the tibioperoneal vessels
  17. Known hypersensitivity or contraindication to nickel-titanium alloy (Nitinol)
  18. Participating in another ongoing investigational clinical trial that has not completed its primary endpoint
  19. Has other comorbidities that, in the opinion of the investigator, would preclude them from receiving this treatment and/or participating in study-required follow-up assessments
  20. Known hypersensitivity or allergy to contrast agents that cannot be medically managed
  21. Thrombolysis of the target vessel within 72 hours prior to the index procedure, where complete resolution of the thrombus was not achieved

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William A. Gray, MD, Principal Investigator — Main Line Health/Lankenau Heart Institute
Locations (39):
- United States (36):
  - Yuma Regional Medical Center, Yuma, Arizona
  - Central Arkansas Veteran's Healthcare System, Little Rock, Arkansas
  - Cedars Sinai Medical Center, Beverly Hills, California
  - Mission Cardiovascular Research Institute, Fremont, California
  - St. Joseph Hospital, Orange, California
  - Denver VA Medical Center, Denver, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Florida Research Network, LLC, Gainesville, Florida
  - Alexian Brothers Medical Center Heart & Vascular Institute, Elk Grove Village, Illinois
  - Adventist Midwest Health, LaGrange, Illinois
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Metro Health Hospital, Wyoming, Michigan
  - Holy Name Medical Center, Teaneck, New Jersey
  - New Mexico Heart Institute, PA, Albuquerque, New Mexico
  - NC Heart and Vascular Research, Raleigh, North Carolina
  - NC Heart and Vascular Research - WakeMed Raleigh, Raleigh, North Carolina
  - Ohio Health Research Institute, Columbus, Ohio
  - Holy Spirit Cardiology, Camp Hill, Pennsylvania
  - St. Mary Medical Center, Langhorne, Pennsylvania
  - Einstein Medical Center Philadelphia, Philadelphia, Pennsylvania
  - Pinnacle Health Cardiovascular Institute, Wormleysburg, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - North Central Heart, Sioux Falls, South Dakota
  - Wellmont CVA Heart Institute, Kingsport, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - North Dallas Research Associates, McKinney, Texas
  - Mission Research Institute, New Braunfels, Texas
  - Sentara Vascular Specialists, Norfolk, Virginia
- Austria (2):
  - Medical University Hospital Graz, Graz
  - Hanusch Krankenhaus, Vienna
- St. Antonius Hospital, Nieuwegein, Utrecht, Netherlands

RESULTS

PARTICIPANT FLOW:
Groups:
- Tack Endovascular System (6F): Use of the Tack Endovascular System (6F) in the superficial femoral and proximal popliteal arteries ranging in diameter from 2.5mm to 6.0mm for the repair of post percutaneous transluminal balloon angioplasty (PTA) dissection(s).
Period: Overall Study
Arm/Group | Tack Endovascular System (6F)
Started | 213 (Intent to Treat (ITT) population.)
Completed | 195 (Completed 12-month follow-up.)
Not Completed | 18
Not completed — Withdrawal by Subject | 6
Not completed — Death | 3
Not completed — Missed 12-month Follow-up | 9

BASELINE CHARACTERISTICS:
Arm/Group | Tack Endovascular System (6F)
Number analyzed (Participants) | 213
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 151
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 195
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 29
  White | 181
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Austria | 40
  United States | 173
BMI [Mean (Standard Deviation); unit: Kg/m^2] — Population: BMI is missing for one subject.
  Kg/m^2
    number analyzed (Participants) | 212
    (all) | 29.3 (6.1)
BMI less than or equal to 30 [Count of Participants; unit: Participants] — Population: BMI is missing for one subject.
  Participants
    number analyzed (Participants) | 212
    (all) | 83
Ankle-brachial index (ABI) in treated leg [Mean (Standard Deviation); unit: ratio] — The ratio of systolic blood pressure measured at the ankle to systolic blood pressure measured at the brachial artery in the arm. Population: ABI information is missing for some subjects
  ratio
    number analyzed (Participants) | 200
    (all) | 0.76 (0.21)
ABI in contralateral limb [Mean (Standard Deviation); unit: ratio] — The ratio of systolic blood pressure measured at the ankle to systolic blood pressure measured at the brachial artery in the arm. ABI was measured in the contralateral (non-treated) limb for comparison to ABI in the treated limb. Population: ABI in contralateral limb is missing for some subjects
  ratio
    number analyzed (Participants) | 190
    (all) | 0.90 (0.18)
Rutherford Classification [Number; unit: participants] — Clinical scale identifying three grades of claudication and three grades of critical limb ischemia. Rutherford Classification ranges from 0 (asymptomatic), 1 (mild claudication), 2 (moderate calcification), 3 (severe calcification), 4 (ischemic rest pain), 5 (minor tissue loss) to 6 (ulceration or gangrene).
  participants
    2 | 68
    3 | 136
    4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Efficacy - Number of Subjects That Met Primary Patency Criteria at 12 Months
Description: Primary patency defined as freedom from Clinical Events Committee (CEC) adjudicated clinically-driven target lesion revascularization (CD-TLR) and freedom from core lab adjudicated duplex ultrasound derived binary restenosis at 12 months (defined as peak systolic velocity ratio (PSVR) >2.5)
Time Frame: 12 Months
Population: ITT population with available data for this assessment.
Measure: Count of Participants; unit: Participants
Groups:
- Tack Endovascular System (6F): Use of the study device in the superficial femoral and/or proximal popliteal arteries ranging in diameter from 2.5mm to 6.0mm for the repair of post percutaneous transluminal balloon angioplasty (PTA) dissection(s)
Arm/Group | Tack Endovascular System (6F)
Number analyzed (Participants) | 183
Participants | 120

2. Primary Outcome: Safety - Number of Subjects That Met the Primary Safety Criteria of Freedom From Major Adverse Events at 30 Days
Description: Freedom from the occurrence of any new-onset major adverse event(s) (MAEs) defined as index limb amputation (above the ankle), CEC adjudicated clinically-driven target lesion revascularization (CD-TLR), or all-cause death at 30 days.
Time Frame: 30 Days
Population: ITT population with available data for this assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Tack Endovascular System (6F)
Number analyzed (Participants) | 212
Participants | 212

ADVERSE EVENTS:
Time Frame: Summary of adverse events that have been reported through 390 days
Arm/Group | Tack Endovascular System (6F)
All-Cause Mortality (participants affected / at risk) | 4/213
Serious Adverse Events (participants affected / at risk) | 115/213
Other Adverse Events (participants affected / at risk) | 139/213
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tack Endovascular System (6F) (N=213)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Anemia aggravated (Blood and lymphatic system disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 3 (3)
Aortic valve stenosis (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Atrial fibrillation with rapid ventricular response (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 2 (2)
Cardiopulmonary arrest (Cardiac disorders) | 1 (1)
Congestive cardiac failure aggravated (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (2)
Non ST segment elevation acute coronary syndrome (Cardiac disorders) | 3 (4)
Non ST segment elevation myocardial infarction (Cardiac disorders) | 2 (2)
Non STEMI (Cardiac disorders) | 1 (1)
Persistent atrial fibrillation (Cardiac disorders) | 1 (1)
Right coronary artery stenosis (Cardiac disorders) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 2 (2)
Unstable angina (Cardiac disorders) | 4 (7)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (3)
Wenckebach (Cardiac disorders) | 1 (1)
Cataract (Eye disorders) | 2 (2)
Double vision (Eye disorders) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
Visual impairment (Eye disorders) | 1 (1)
Acute pancreatitis (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Diarrhea recurrent (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Esophageal varices (Gastrointestinal disorders) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 1 (1)
Gastroparesis (Gastrointestinal disorders) | 1 (1)
Hernia abdominal wall (Gastrointestinal disorders) | 1 (1)
Pain epigastric (Gastrointestinal disorders) | 1 (1)
Rectal bleeding (Gastrointestinal disorders) | 1 (1)
Right inguinal hernia (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal bleeding (Gastrointestinal disorders) | 2 (2)
Chest pain (General disorders) | 4 (5)
Chest pressure (General disorders) | 1 (1)
Edema (General disorders) | 1 (1)
Medical device site thrombosis (General disorders) | 2 (2)
Pain worsened (General disorders) | 1 (1)
Peripheral edema (General disorders) | 1 (1)
Swelling of feet (General disorders) | 1 (1)
Swelling of legs (General disorders) | 1 (1)
Weakness (General disorders) | 1 (1)
Acute cholecystitis (Hepatobiliary disorders) | 1 (1)
Gallbladder sludge (Hepatobiliary disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Anaphylaxis (Immune system disorders) | 1 (1)
Acute bronchitis (Infections and infestations) | 1 (1)
Acute diverticulitis (Infections and infestations) | 1 (1)
Acute osteomyelitis (Infections and infestations) | 1 (1)
Cellulitis of toe (Infections and infestations) | 1 (1)
Diarrhea, Clostridium difficile (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Influenza B virus infection (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Osteomyelitis acute (Infections and infestations) | 1 (1)
Pneumonia, organism unspecified (Infections and infestations) | 5 (5)
Pyelonephritis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection, site not specified (Infections and infestations) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Nausea postoperative (Injury, poisoning and procedural complications) | 1 (1)
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 17 (20)
Post embolization syndrome (Injury, poisoning and procedural complications) | 3 (3)
Post procedural hematoma (Injury, poisoning and procedural complications) | 2 (2)
Subdural hematoma (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm ruptured (Injury, poisoning and procedural complications) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cervical disc herniation (Musculoskeletal and connective tissue disorders) | 1 (1)
Cervical pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Ganglion cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Groin discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal stenosis of lumbar region (Musculoskeletal and connective tissue disorders) | 1 (1)
Glomus tympanicum tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carotid artery disease (Nervous system disorders) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 3 (4)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1)
Lumboischialgia (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Neurogenic bladder (Renal and urinary disorders) | 1 (1)
Stone urinary bladder (Renal and urinary disorders) | 1 (1)
COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Chronic obstructive lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Accelerated hypertension (Vascular disorders) | 1 (1)
Arteriovenous fistula, acquired (Vascular disorders) | 1 (1)
Claudication (Vascular disorders) | 23 (31)
Critical limb ischemia (Vascular disorders) | 4 (4)
Femoral artery occlusion (Vascular disorders) | 3 (3)
Femoral artery stenosis (Vascular disorders) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1)
Iliac artery stenosis (Vascular disorders) | 1 (1)
Melena (Vascular disorders) | 1 (1)
Peripheral arterial disease (Vascular disorders) | 9 (9)
Peripheral artery dissection (Vascular disorders) | 2 (2)
Peripheral artery occlusion (Vascular disorders) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1)
Peripheral vascular disease (Vascular disorders) | 9 (11)
Popliteal arterial stenosis (Vascular disorders) | 1 (1)
Popliteal stenosis (Vascular disorders) | 1 (1)
Superficial femoral arterial stenosis (Vascular disorders) | 1 (1)
Thrombosis of leg deep venous (Vascular disorders) | 1 (1)
Uncontrolled hypertension (Vascular disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tack Endovascular System (6F) (N=213)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Anemia aggravated (Blood and lymphatic system disorders) | 1 (1)
Anemia iron deficiency (Blood and lymphatic system disorders) | 1 (1)
Anemia post chemotherapy (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 3 (3)
Angina pectoris aggravated (Cardiac disorders) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Atrial fibrillation with rapid ventricular response (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Cardiopulmonary arrest (Cardiac disorders) | 1 (1)
Congestive cardiac failure aggravated (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 3 (3)
Coronary artery disease progression (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 3 (3)
Left bundle branch block (Cardiac disorders) | 1 (1)
Non ST segment elevation acute coronary syndrome (Cardiac disorders) | 3 (4)
Non ST segment elevation myocardial infarction (Cardiac disorders) | 3 (3)
Non STEMI (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Paroxysmal atrial fibrillation (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Persistent atrial fibrillation (Cardiac disorders) | 1 (1)
Recurrent atrial fibrillation (Cardiac disorders) | 1 (1)
Right coronary artery stenosis (Cardiac disorders) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Unstable angina (Cardiac disorders) | 4 (7)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (3)
Wenckebach (Cardiac disorders) | 1 (1)
Cystic kidney disease (Congenital, familial and genetic disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Earache (Ear and labyrinth disorders) | 1 (1)
Sensation of pressure in ear (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Goiter (Endocrine disorders) | 1 (1)
Cataract (Eye disorders) | 2 (2)
Cataract (left) (Eye disorders) | 1 (1)
Diabetic macular edema (Eye disorders) | 1 (1)
Double vision (Eye disorders) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
Visual impairment (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Acute pancreatitis (Gastrointestinal disorders) | 1 (1)
Appendix disorder (Gastrointestinal disorders) | 1 (1)
Bilateral inguinal hernia (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dental disorder NOS (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Diarrhea recurrent (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Esophageal spasm (Gastrointestinal disorders) | 1 (1)
Esophageal varices (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 1 (1)
Gastroparesis (Gastrointestinal disorders) | 1 (1)
Hernia abdominal wall (Gastrointestinal disorders) | 1 (1)
Pain epigastric (Gastrointestinal disorders) | 1 (1)
Rectal bleeding (Gastrointestinal disorders) | 1 (1)
Retroperitoneal bleeding (Gastrointestinal disorders) | 1 (1)
Right inguinal hernia (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal bleeding (Gastrointestinal disorders) | 2 (2)
Adverse drug reaction (General disorders) | 1 (1)
Chest pain (General disorders) | 8 (9)
Chest pressure (General disorders) | 1 (1)
Chronic edema of legs (General disorders) | 1 (1)
Complication of device insertion (General disorders) | 1 (1)
Device failure (General disorders) | 1 (1)
Drug side effect (General disorders) | 1 (1)
Edema (General disorders) | 1 (1)
Leg edema (General disorders) | 2 (2)
Medical device site thrombosis (General disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Pain chest (General disorders) | 1 (1)
Pain worsened (General disorders) | 1 (1)
Peripheral edema (General disorders) | 1 (1)
Swelling of feet (General disorders) | 1 (1)
Swelling of legs (General disorders) | 1 (1)
Unevaluable event (General disorders) | 1 (1)
Weakness (General disorders) | 1 (1)
Acute cholecystitis (Hepatobiliary disorders) | 1 (1)
Gallbladder sludge (Hepatobiliary disorders) | 1 (1)
Hepatic cyst (Hepatobiliary disorders) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1)
Liver cirrhosis (Hepatobiliary disorders) | 1 (1)
Steatosis hepatic (Hepatobiliary disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 2 (2)
Anaphylaxis (Immune system disorders) | 1 (1)
Acute bronchitis (Infections and infestations) | 3 (3)
Acute diverticulitis (Infections and infestations) | 1 (1)
Acute osteomyelitis (Infections and infestations) | 1 (1)
Cellulitis of foot (Infections and infestations) | 1 (1)
Cellulitis of leg (Infections and infestations) | 2 (2)
Cellulitis of toe (Infections and infestations) | 1 (1)
Cold (Infections and infestations) | 1 (1)
Common cold (Infections and infestations) | 3 (3)
Diarrhea, Clostridium difficile (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1)
Foot infection (Infections and infestations) | 1 (1)
Hepatitis C (Infections and infestations) | 1 (1)
Influenza B virus infection (Infections and infestations) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1)
Lyme disease (Infections and infestations) | 1 (1)
Nasal abscess (Infections and infestations) | 1 (1)
Onychomycosis (Infections and infestations) | 1 (2)
Osteomyelitis (Infections and infestations) | 1 (1)
Osteomyelitis acute (Infections and infestations) | 1 (1)
Pneumonia, organism unspecified (Infections and infestations) | 6 (6)
Pyelonephritis (Infections and infestations) | 1 (1)
Respiratory infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Shingles (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection aggravated (Infections and infestations) | 1 (1)
Tinea pedis (Infections and infestations) | 1 (1)
Urinary tract infection, site not specified (Infections and infestations) | 3 (3)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 3 (3)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (3)
Laceration of hand (Injury, poisoning and procedural complications) | 1 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1)
Nausea postoperative (Injury, poisoning and procedural complications) | 1 (1)
Open wound of fingers, without mention of complication (Injury, poisoning and procedural complications) | 1 (1)
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 18 (22)
Post embolization syndrome (Injury, poisoning and procedural complications) | 3 (3)
Post procedural hematoma (Injury, poisoning and procedural complications) | 9 (9)
Spider bite (Injury, poisoning and procedural complications) | 1 (1)
Stress fracture (Injury, poisoning and procedural complications) | 1 (1)
Subdural hematoma (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm ruptured (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 2 (2)
Blood sugar increased (Investigations) | 1 (1)
Folic acid deficiency (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypoglycemia, unspecified (Metabolism and nutrition disorders) | 1 (1)
Osteoporosis (Metabolism and nutrition disorders) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1)
Arthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Back pain aggravated (Musculoskeletal and connective tissue disorders) | 2 (2)
Calf pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cervical disc herniation (Musculoskeletal and connective tissue disorders) | 1 (1)
Cervical pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Degeneration of lumbar or lumbosacral intervertebral disc (Musculoskeletal and connective tissue disorders) | 1 (1)
Foot pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Ganglion cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Gonarthrosis (Musculoskeletal and connective tissue disorders) | 3 (3)
Groin discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Herniated disc (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc bulging (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Leg pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Low back pain (Musculoskeletal and connective tissue disorders) | 1 (3)
Lower extremities weakness of (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in hip (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Prolapsed lumbar disc (Musculoskeletal and connective tissue disorders) | 1 (1)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal stenosis of lumbar region (Musculoskeletal and connective tissue disorders) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Glomus tympanicum tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Mucinous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Burning sensation (Nervous system disorders) | 1 (3)
Carotid artery disease (Nervous system disorders) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 3 (4)
Carpal tunnel syndrome (Nervous system disorders) | 1 (2)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Headache aggravated (Nervous system disorders) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1)
Lumboischialgia (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Numbness in feet (Nervous system disorders) | 2 (3)
Numbness of extremities (Nervous system disorders) | 1 (1)
Restless legs (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
TIA (Nervous system disorders) | 1 (1)
Tension headache (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (3)
Hematuria (Renal and urinary disorders) | 1 (1)
Neurogenic bladder (Renal and urinary disorders) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1)
Stone urinary bladder (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Epididymal cyst (Reproductive system and breast disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Prostatic hypertrophy (Reproductive system and breast disorders) | 2 (2)
Vaginal bleeding (Reproductive system and breast disorders) | 1 (1)
Bleeding nose (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
COPD (Respiratory, thoracic and mediastinal disorders) | 2 (2)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Chronic obstructive lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Exertional dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung nodule (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1)
Facial swelling (Skin and subcutaneous tissue disorders) | 1 (1)
Foot callus (Skin and subcutaneous tissue disorders) | 1 (1)
Heel ulcer (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Accelerated hypertension (Vascular disorders) | 1 (1)
Arterial perforation (Vascular disorders) | 1 (1)
Arterial thrombosis limb (Vascular disorders) | 2 (2)
Arteriovenous fistula, acquired (Vascular disorders) | 1 (1)
Bleeding (Vascular disorders) | 1 (1)
Chronic venous insufficiency (Vascular disorders) | 1 (1)
Claudication (Vascular disorders) | 28 (37)
Critical limb ischemia (Vascular disorders) | 4 (4)
Dry gangrene (Vascular disorders) | 1 (1)
Femoral artery dissection (Vascular disorders) | 1 (1)
Femoral artery occlusion (Vascular disorders) | 4 (4)
Femoral artery stenosis (Vascular disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hypertension aggravated (Vascular disorders) | 1 (1)
Hypertension worsened (Vascular disorders) | 4 (4)
Hypertensive crisis (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Iliac artery dissection (Vascular disorders) | 1 (1)
Iliac artery stenosis (Vascular disorders) | 1 (1)
Intermittent claudication (Vascular disorders) | 1 (1)
Lymphedema (Vascular disorders) | 1 (1)
Melena (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Peripheral arterial disease (Vascular disorders) | 11 (11)
Peripheral artery dissection (Vascular disorders) | 4 (4)
Peripheral artery occlusion (Vascular disorders) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1)
Peripheral vascular disease (Vascular disorders) | 11 (13)
Popliteal arterial stenosis (Vascular disorders) | 1 (1)
Popliteal stenosis (Vascular disorders) | 1 (1)
Posterior tibial artery perforation (Vascular disorders) | 1 (1)
Superficial femoral arterial stenosis (Vascular disorders) | 1 (1)
Thrombosis of leg deep venous (Vascular disorders) | 1 (1)
Uncontrolled hypertension (Vascular disorders) | 1 (1)
Varicose veins (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI acknowledges that Clinical Trial is part of multi-center clinical study. Publication of multi-center data requires prior review and consent of both Sponsor and all participating sites. PI agrees that the first publication of the results of the Clinical Trial shall be made in conjunction with results from other participating sites. Provided, however, that if no multi-center publication is made within one year from database lock, then PI may publish individually.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-10): https://cdn.clinicaltrials.gov/large-docs/84/NCT02522884/Prot_SAP_000.pdf